CLINICAL TRIAL: NCT04315922
Title: Multiomics Targeting Microbiome Associated Changes in Stroke Patients (StrokeMicroBiomics)
Acronym: SMB
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University of Luxembourg (Other)
Responsible Party: Principal Investigator, Philip William Melton, MD, Ludwig-Maximilians - University of Munich
Other Study IDs: Synergy ID 390857198 SMB
Record Dates: First submitted 2020-03-12; First posted 2020-03-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: Microbiome; Immune System; Metabolome; Brain Lesion; Gut-Brain Axis
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and blood samples collected at both acute and chronic timepoints from study participants are stored at -80°C in on-site Biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe Ischemic Stroke: Severe Stroke as defined by inclusion criteria
  Interventions: Diagnostic Test: Microbiome and Plasma Characterisation
- Mild Ischemic Stroke: Mild Stroke as defined by inclusion criteria
  Interventions: Diagnostic Test: Microbiome and Plasma Characterisation
- Transient Ischemic Attack: Transient Ischemic Attack as defined by inclusion criteria
  Interventions: Diagnostic Test: Microbiome and Plasma Characterisation

INTERVENTIONS:
Diagnostic Test: Microbiome and Plasma Characterisation — Flow Cytometry, Mass-Spectometry, Shotgun-Sequencing

SUMMARY:
Preclinical research has established a convincing connection between changes in the gut microbiota composition and stroke outcome. However clinical data on the gut-brain axis, and its chronic characteristics, is sparse. Additional investigations in the context of ischemic stroke regarding the relationship between dysbiosis and functional changes of the microbiome, as characterized by the metabolome, are still required. The StrokeMicroBiomics study will offer insight into these mechanisms and offer new potential targets for therapeutic interventions.

The primary objective is the characterisation of gut dysbiosis in ischemic stroke patients in the acute phase after stroke and during a 3 month follow-up period.

The secondary objectives include the identification of dysregulated gut microbiome metabolites and key immune cell populations in addition to the clinical progression of the study participants during the 3 month follow-up period after disease onset.

DETAILED DESCRIPTION:
Results of experimental, preclinical studies suggest that microbiome-targeted may improve stroke outcome as well as stroke-related comorbidities. Yet, clinical trials describing the extent and time course of microbiome changes after stroke are currently not available. Moreover, the impact of post-stroke dysbiosis on metabolic changes and the systemic immunity are unexplored.

Therefore, the primary objective of this trial is the characterization of gut dysbiosis progression in ischemic stroke patients during a 3 month follow-up period .

The secondary objectives include the identification of dysregulated gut microbiome metabolites and key immune cell populations in addition to the clinical progression of the study participants during the 3 month follow-up period after disease onset.

In order to elucidate the differential impact of lesion size on immune and microbiome homeostasis, separate patient cohorts with mild and severe stroke will be studied.

Furthermore, to control for the effects of temporary focal neurological deficits and stress induced microbiome and immune changes, patients with stroke mimics and transient ischemic attacks (TIA) are being recruited to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Written consent as submitted and approved to the human subjects review board must be gathered from the participants
* Participants must be at least 50 years of age

For the severe stroke cohort, eligibility is defined by:

* CT or MRI confirmed ischemic stroke affecting at least 1/3 of the anterior, medial or posterior cerebral arteries cortical coverage
* NIHSS of at least 10 at time of induction into emergency room
* Ischemic Stroke occured within the last 7 days

For the mild stroke cohort, eligibility is defined by:

* CT or MRI confirmed ischemic stroke affecting no more than 1/3 of the anterior, medial or posterior cerebral arteries cortical coverage
* NIHSS between 1 and 10 at time of induction into emergency room
* Ischemic Stroke occured within the last 7 days

For the TIA cohort, eligibility is defined by:

* CT or MRI confirmed absence of a lesion
* NIHSS of 0 no more than 24 hours after induction into emergency room
* TIA occured within the last 7 days

Exclusion Criteria:

* Pregnancy
* Diagnosed and malignant Tumor ailment
* Active, non-stroke related immunosuppression (i.e. HIV)
* Infection, operative procedure or antibiotics treatment within 4 weeks prior to stroke/TIA
* Relevant autoimmune disease (i.e Morbus Crohn)
* Chronic infectious diseases (i.e Hepatitis C)
* Hemorrhagic Stroke or intracranial bleeding
* Cerebellar lesions
* Other neurodegenerative diseases (i.e. Parkinson´s Disease or Alzheimers Dementia)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are recruited and samples taken within 7 days of either stroke or TIA onset.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in the Gut Microbiome Composition at 3 Months post Stroke/TIA | 1-7 Days and 90 Days after Stroke
  Gut Microbiome Composition is assessed using Shotgun Sequencing
Changes from Baseline of the Gut Metabolome as measured in Blood and Stool at 3 Months post Stroke/TIA | 1-7 Days and 90 Days after Stroke
  The Metabolome is measured using Mass-Spectometry
Changes from Baseline in key Immune Populations at 3 Months post Stroke/TIA | 1-7 Days and 90 Days after Stroke
  Immune Populations are measured using Flow Cytometry

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | 1-7 days and 90 days after stroke
Modified Rankin Score (mRS) | 1-7 days and 90 days after stroke
CT and (if available) MRI documentation | 1-7 days and 90 days after stroke

CONTACTS AND LOCATIONS:
Locations (1):
- LMU University hospital, Munich, Munich, Bavaria, Germany